CLINICAL TRIAL: NCT04591873
Title: Application of Telemedicine to Optimize Teamwork and Infection Control of Critical Patients in Isolation Rooms in the Emergency Department During Novel Coronavirus Disease 2019 Outbreak
Brief Title: Using Telemedicine to Optimize Teamwork and Infection Control of Critical and Highly-infectious Patients in an Emergency Department
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202007114RINA
Record Dates: First submitted 2020-09-23; First posted 2020-10-19 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2020-10

CONDITIONS: Critical Illness; Infections, Respiratory; Emergency Service, Hospital; Telemedicine
Keywords: telemedicine; isolation; critical care; emergency medicine; COVID-19
MeSH Terms: conditions — Critical Illness; Respiratory Tract Infections; Emergencies; COVID-19 | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critical patients in the emergency department
  Interventions: Other: telemedicine; Other: traditional communication tools

INTERVENTIONS:
Other: telemedicine — Using telemedicine system to communicate
Other: traditional communication tools — Use telephone or direct verbal communication

SUMMARY:
Since 2000, various emerging infectious diseases have repeatedly caused serious impact on the health of the global population and the healthcare systems. With the growing international transportation and improving accessibility of the healthcare systems, hospitals have been inevitably the first sentinels dealing with emerging infectious diseases. The biological disasters, such as the Severe Acute Respiratory Syndrome (SARS) in 2003, the Middle East Respiratory Syndrome (MERS) outbreak in South Korean in 2015, and the Coronavirus disease 2019 (COVID-19) outbreak this year, challenged our vulnerable healthcare systems and caused great loss of lives.

Regarding the ongoing global epidemics and possible community outbreaks of the COVID-19, the management of biological disasters for an overcrowded emergency department should be planned. In the early 2020, the emergency department used a double-triage and telemedicine method to treat non-critical patient with suspected COVID-19. This application reduced the exposure time of the first responders and reserve adequate interview quality. However, for the critical patients treated in the isolated resuscitation rooms, the unique environment limited the teamwork and communication for the resuscitation team. These factors might led to poorer quality of critical care.

The investigators designed a telemedicine-teamwork model, which connected the isolation room, prepare room and nursing station by an video-conferencing system in the emergency department. This model try to break the barriers of space between the rooms and facilitate the teamwork communications between each unit. Besides, by providing a more efficient workflow, this model could lower the total exposure time for all workers in the contaminated area. This study was conducted to evaluate the benefits of the telemedicine-teamwork model and provide a practical, safe and effective alternative to critical care of the patients with suspected highly infectious diseases.

ELIGIBILITY:
For patients:

1.Patients triaged as highly-infectious patients, needed to be treated in isolation rooms in the emergency department.

For healthcare providers:

1. Those providers who participates in the critical care for the patients included in the study accordingly

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients triaged as highly-infectious patients, needed to be treated in isolation rooms in the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
time to complete intubation | immediately after intervention

SECONDARY OUTCOMES:
teamwork score | immediately after intervention
  Team Emergency Assessment Measure, minimal score is 0 and the maximal score is 4. Higher score means a better outcome.
exposure time in isolation rooms | immediately after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hao Lin, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lin CH, Lin HY, Wu SN, Tseng WP, Chen WT, Tien YT, Wu CY, Huang CH, Tsai MS. Using a telemedicine-assisted airway model to improve the communication and teamwork of tracheal intubation during the coronavirus disease 2019 pandemic. J Telemed Telecare. 2024 Aug;30(7):1140-1148. doi: 10.1177/1357633X221124175. Epub 2022 Sep 6. PMID 36066025